CLINICAL TRIAL: NCT03291691
Title: The Use of Protective Nerve Stimulation in Different Regional Anesthetic Blocks (Interscalene, Axillary, Femoral and Sciatic Nerve Blocks)
Brief Title: Protective Nerve Stimulation in Regional Anesthesia
Acronym: ProNerv
Status: Suspended | Type: Observational
Why Stopped: for organizational reasons
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jurgen Birnbaum, Principal Investigator and Consultant of the Department of Anesthesiology and Operative Intensive Care Medicine, CCM and CVK, Charite University, Berlin, Germany
Other Study IDs: ProNerv
Record Dates: First submitted 2017-07-25; First posted 2017-09-25 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia, Local; Nerve Block; Brachial Plexus Block
Keywords: Protective Nerve Stimulation; Regional Anesthesia; Sciatic nerve block; femoral nerve block; brachial plexus block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Standard of care: SCI: Patients at Charite, with lower limb surgery undergoing a protective performed ultrasound guided sciatic nerve block. N=15.
- Standard of care: FEM: Patients at Charite, with lower limb surgery undergoing a protective performed ultrasound guided femoral nerve block. N=15.
- Standard of care: ISB: Patients at Charite, with upper limb surgery undergoing a protective performed ultrasound guided interscalene plexus block. N=15.
- Standard of care: AXP: Patients at Charite, with upper limb surgery undergoing a protective performed ultrasound guided axillary plexus block. N=15.

SUMMARY:
Peripheral nerve blocks can be conducted with ultrasound, electrical nerve stimulation or landmark technique or a combination of this techniques. Whether a regional block should be conducted with a combination of those different possibilities is highly discussed. In this study the investigators want to show the effectiveness of new standard way of combined use of ultrasound and nerve stimulation, they call protective nerve stimulation. According to ethical vote we are conducting an observational study.

DETAILED DESCRIPTION:
All patients will get the regional block they need for the elective surgery. Before starting the block a standard monitoring will be established. After applying the monitoring the block will be performed by an experienced anesthetist in supervision of another experienced anesthetist. The nerve stimulator is set on a fixed current of 1.0 mA and a block without motoric response on this current is tried. Ultrasound images are saved. After performing the regional anesthesia the further anesthetic procedure will be carried out and the surgery will take place. After surgery the patients will be transported to the recovery room or Postanesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age of 18 or older
* elective surgery patients at Campus Charité Mitte with clinical benefit of regional anesthesia

Exclusion Criteria:

* existing contraindication for regional nerve blocks or the use of Protective Nerve Stimulation
* patients who undergo outpatient treatment
* allergy against local anesthetics
* age under 18 years
* Lacking willingness to take part in the study
* ASA PS score of 4 or more
* preexisting neural damage in the effect area
* Diabetes mellitus, alcohol use disorder
* Participation in other prospective clinical interventional trials
* Accommodation in an institution due to an official or judicial order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 female and male patients undergoing elective surgery with a regional block at Charité -Universitätsmedizin Berlin
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectivity | Duration of preparation, surgery and recovery room (an average of 4 hours)
  Effective motor blockade and sensitive blockade at fixed timepoints

SECONDARY OUTCOMES:
Muscle contractions | Duration of preparation, surgery and recovery room (an average of 4 hours)
  Number of expected and unexpected muscle contractions
Paresthesia | Duration of preparation, surgery and recovery room (an average of 4 hours)
  Number of expected and unexpected paresthesia
Pain while blocking | Duration of preparation, surgery and recovery room (an average of 4 hours)
  Does the patient have pain while blocking? Pain during hospital stay will be measured with the Numeric Rating Scale (NRS-V). For patients unable of pain self-assessment (e.g. ventilated patients, patients in delirious state or patients with stroke affecting language skills) observer-rated pain scales will be applied: Behavioural Pain Scale (BPS for ventilated) and BPS-NI (for non-ventilated) patients.
Pain after surgery | Duration of preparation, surgery and recovery room (an average of 4 hours)
  Does the patient have pain after surgery? Pain during hospital stay will be measured with the Numeric Rating Scale (NRS-V). For patients unable of pain self-assessment (e.g. ventilated patients, patients in delirious state or patients with stroke affecting language skills) observer-rated pain scales will be applied: Behavioural Pain Scale (BPS for ventilated) and BPS-NI (for non-ventilated) patients.
Satisfaction | Duration of preparation, surgery and recovery room (an average of 4 hours)
  Satisfaction of the patient in a 6-step Likert scale
Impedance | Duration of preparation, surgery and recovery room (an average of 4 hours)
  impedance measured by the nerve stimulator while proceeding with the needle
Changes of impedance | Duration of preparation, surgery and recovery room (an average of 4 hours)
  changes of impedance measured by the nerve stimulator while proceeding with the needle

OTHER OUTCOMES:
Bloody Tap | Duration of preparation, surgery and recovery room (an average of 4 hours)
  Appearance of Bloody Tap before, during and after the block (yes/no)
Postoperative Nausea and Vomiting | Duration of preparation, surgery and recovery room (an average of 4 hours)
  Appearance of PONV before, during and after the block (yes/no)
pruritus | Duration of preparation, surgery and recovery room (an average of 4 hours)
  Appearance of pruritus before, during and after the block (yes/no)
Analgetics consumption | Duration of preparation, surgery and recovery room (an average of 4 hours)
  Amount of opioids needed before, during and after the surgery until the patient leaves the recovery unit

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Birnbaum, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin Campus Charité Mitte, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salem MH, Winckelmann J, Geiger P, Mehrkens HH, Salem KH. Electrostimulation with or without ultrasound-guidance in interscalene brachial plexus block for shoulder surgery. J Anesth. 2012 Aug;26(4):610-3. doi: 10.1007/s00540-012-1366-x. Epub 2012 Mar 4. PMID 22391670
- [Background] Klaastad O, Sauter AR, Dodgson MS. Brachial plexus block with or without ultrasound guidance. Curr Opin Anaesthesiol. 2009 Oct;22(5):655-60. doi: 10.1097/ACO.0b013e32832eb7d3. PMID 19550303
- [Background] Dillane D, Tsui BC. Is there still a place for the use of nerve stimulation? Paediatr Anaesth. 2012 Jan;22(1):102-8. doi: 10.1111/j.1460-9592.2011.03729.x. Epub 2011 Nov 4. PMID 22050512
- [Background] Vassiliou T, Muller HH, Limberg S, De Andres J, Steinfeldt T, Wiesmann T. Risk evaluation for needle-nerve contact related to electrical nerve stimulation in a porcine model. Acta Anaesthesiol Scand. 2016 Mar;60(3):400-6. doi: 10.1111/aas.12664. Epub 2015 Dec 15. PMID 26666693
- [Background] Dexter F, Candiotti KA. Multicenter assessment of the Iowa Satisfaction with Anesthesia Scale, an instrument that measures patient satisfaction with monitored anesthesia care. Anesth Analg. 2011 Aug;113(2):364-8. doi: 10.1213/ANE.0b013e318217f804. Epub 2011 Apr 25. PMID 21519043
- [Background] Wiesmann T, Borntrager A, Vassiliou T, Hadzic A, Wulf H, Muller HH, Steinfeldt T. Minimal current intensity to elicit an evoked motor response cannot discern between needle-nerve contact and intraneural needle insertion. Anesth Analg. 2014 Mar;118(3):681-6. doi: 10.1213/ANE.0b013e3182a94454. PMID 24284806
- [Background] Wiesmann T, Steinfeldt T, Exner M, Nimphius W, De Andres J, Wulf H, Schwemmer U. Intraneural injection of a test dose of local anesthetic in peripheral nerves - does it induce histological changes in nerve tissue? Acta Anaesthesiol Scand. 2017 Jan;61(1):91-98. doi: 10.1111/aas.12825. Epub 2016 Oct 25. PMID 27778324
- [Background] Sen O, Sayilgan NC, Tutuncu AC, Bakan M, Koksal GM, Oz H. Evaluation of sciatic nerve damage following intraneural injection of bupivacaine, levobupivacaine and lidocaine in rats. Braz J Anesthesiol. 2016 May-Jun;66(3):272-5. doi: 10.1016/j.bjane.2014.09.012. Epub 2015 Mar 12. PMID 27108824
- [Background] Brull R, McCartney CJ, Chan VW, El-Beheiry H. Neurological complications after regional anesthesia: contemporary estimates of risk. Anesth Analg. 2007 Apr;104(4):965-74. doi: 10.1213/01.ane.0000258740.17193.ec. PMID 17377115